CLINICAL TRIAL: NCT03249038
Title: Estimated Blood Loss: Novel Model for Estimating Surgical Blood Loss.
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Sebastian Jaramillo, Dr. Sebastian Jaramillo, Hospital Clinic of Barcelona
Other Study IDs: HCB/2016/0906
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Blood Loss, Surgical; Blood Loss; Blood Loss, Postoperative
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage; Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Serum hemoglobin concentration.
  * Hemoglobin concentration of external blood loss.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of external blood loss
Diagnostic Test: Serum Hemoglobin concentration

SUMMARY:
Estimated blood loss is an important parameter recognized as a standard practice in anesthesiology and others medical specialties, with relevant clinical and research applications. Currently is no model capable of accurately estimate blood loss. The purpose of this study is to evaluate the accuracy of a novel model.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective urologic laparoscopy surgery.

Exclusion Criteria:

* Patient with suspected or confirmed heart failure, severe hypertension, hepatic cirrhosis, chronic kidney disease on dialysis, coagulopathy, as well as patient receiving diuretics, anticoagulant or antiplatelet agents.
* Cases in which surgical gauzes were used, including conversion to open surgical technique. - Patients who have received transfusions of RBCs during the perioperative period.
* Patients who have showed postoperative bleeding, defined by an amount greater than 50 ml in surgical drains, or any other type of blood loss.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective urologic laparoscopy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin mass lost | Intraoperative
Postoperative serum hemoglobin concentration | 48 hours

IPD SHARING:
Plan to Share IPD: No